CLINICAL TRIAL: NCT02555111
Title: Multicentric Randomized Study of Xarelto Versus no Treatment for the Prevention of Recurrent Thrombosis in Patients With Chronic Portal Vein Thrombosis.
Brief Title: Xarelto Versus no Treatment for the Prevention of Recurrent Thrombosis in Patients With Chronic Portal Vein Thrombosis.
Acronym: RIPORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM 11077 - P 110150; 2015-001190-40 (EudraCT Number)
Record Dates: First submitted 2015-08-28; First posted 2015-09-21 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2020-03

CONDITIONS: Deep Vein Thrombosis; Chronic Portal Vein Thrombosis
Keywords: thrombosis
MeSH Terms: conditions — Venous Thrombosis; Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xarelto (Experimental): 15mg/day oral administration during 2 to 4 years (based on the recruitment date).
  Interventions: Drug: Xarelto
- untreated (No Intervention): the patient won't receive any treatment during his study participation.

INTERVENTIONS:
Drug: Xarelto — 15mg/day oral administration during 2 to 4 years (based on the recruitment date).
  Other Names: Rivaroxaban
  Arms: Xarelto

SUMMARY:
Open randomized therapeutic study to assess the efficacy of Xarelto 15mg/day in the recurrence of thromboembolic event compared to an untreated group in patients with chronic portal vein thrombosis without high risk thrombophilia.

DETAILED DESCRIPTION:
Chronic portal vein thrombosis (PVT) is a rare disease, affecting young patients, characterized by permanent obstruction of the portal vein trunk causing portal hypertension. In 60-70% of cases it is related to high risk, moderate or mild prothrombotic risk factors.

Accordingly, there are 2 types of complications from PVT :(i) gastrointestinal haemorrhage related to portal hypertension; and (ii) recurrent thrombosis.

Recurrent thrombosis its most dreaded complication as it may lead to intestinal infarction with a related mortality of 20-60% and a high risk of intestinal insufficiency.

Gastrointestinal haemorrhage related to portal hypertension occurs in 20% patients/year. It is less frequent in patients treated with medical or endoscopic prophylaxis for variceal bleeding.

Retrospective data shows that anticoagulation does not worsen the prognosis, and may conversely improve it. Thus, in patients at risk for gastrointestinal bleeding due to portal hypertension and a mild or moderate risk of recurrent thrombosis, the benefit-risk ratio of anticoagulation therapy is unclear.

The aim of this open randomised trial is to assess the efficacy of Xarelto 15mg/day, a new oral factor Xa inhibitor, in the recurrence of thromboembolic event and the risk of major bleeding compared to an untreated group in patients with chronic portal vein thrombosis without high risk thrombophilia.

The hypothesis of the trial is that treatment with Xarelto® would reduce the risk of recurrence of acute deep vein thrombosis (DVT) regardless location, with limited increase in the risk of hemorrhage in patients with chronic portal thrombosis and no high-risk factors for thrombosis recurrence

This is a national, multicentric, interventional study. 17 french centers already agreed to participate.

296 patients will be included on a 3 years period with 2 to 4 years treatment period. All data will be collected after informed consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 18 to 90 years old
* Patients either with :

  * Portal cavernoma radiologically confirmed, treated or not by anticoagulant
  * previous history of acute portal thrombosis for more than 6 months confirmed by angio-TDM or angio-MRI, repermeabilized or not
* prophylaxis of gastro-intestinal bleeding due to portal hypertension, as recommended for cirrhosis patients. Upper gastro-intestinal endoscopy for less than 12 months
* clinical examination
* for women of childbearing age, contraception, either mecanichal or intra-uterin device, or oral progestative alone. No oral oestroprogestative contraception is allowed.
* written informed consent
* covered by a social security scheme or French "CMU"

Exclusion Criteria:

* At least one High risk factors of thrombosis recurrence after review by the committee composed of an hepatologist and an hematologist specialist of hemostasis
* Cirrhosis clinically or histologically confirmed or Budd-Chiari syndrome
* Any disease leading to significant coagulopathy and clinically significant bleeding risk (platelets <50 000, or PT <30% without VKA, or Factor V <30% or Fibrinogen <0,8).
* Personal or familial (1rst degree) history of spontanaeous deep vein thrombosis requiring anticoagulant treatment
* pregnant or breast-feeding women
* History of mesenteric veinous ischemia leading to intestinal resection
* patient infected by HIV and treated by anti-protease
* Formal indication to anticoagulant treatment for any reason
* No possible follow-up
* severe renal injury (creatinin clearance <30 ml/min)
* Patients receiving a systemic treatment by azoled antifongic agent (such as ketoconazole, itraconazole, voriconazole or posaconazole), or a protease inhibitor. These are strong CYP3A4 and P-gp inhibitors.
* Patients receiving a systemic treatment by rifampicyn or any other strong CYP3A4 inducting/stimulator (phenytoïne, carbamazepine, phenobarbital or millepertuis/Hypericum perforatum)
* Hypersensitvity to rivaroxaban or excipients
* active bleeding, or any condition at risk for significant major bleeding
* Any other concomitant anticoagulant treatment, such as non-fractionnaed heparin, low-molecular weight heparin (enoxaparin, dalteparine, etc…), heparin derivatives (fondaparinux, etc), oral anticoagulant (warfarine, dabigatran etexilate, apixaban, etc) except in case of switch to Xarelto® or, in case of non-fractionnaed heparin administered to maintain central veinous or arterial catheterism permeability
* Concomitant treatment by clopidogrel / Plavix® for acute coronary syndrome
* hepatic transplantation
* Intra-hepatic shunt

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Incidence of thromboembolic event in any territory ( splanchnic or extra splanchnic, lower limbs, cerebral veinous thrombosis, pulmonary embolism) or death | 2 years
  In patients with chronic portal vein thrombosis without high risk thrombophilia, to assess the efficacy of Xarelto in the recurrence of thromboembolic event compared to absence of treatment.

SECONDARY OUTCOMES:
Efficacy of xarelto | 2 years
  Assess the efficacy regarding:
  - Incidence of Pulmonary embolism, Deep vein thrombosis, Major bleedings and Portal hypertension bleeding, new non bleeding complication of portal hypertension, minor bleeding,
Safety of xarelto | 2 years
  Assess the safety regarding:
  * Toxicity of Xarelto, especially hepatic.
  * Gastrointestinal clinically relevant non major bleedings related to portal hypertension
  * Other gastrointestinal clinically relevant non major bleedings
  * Other adverse events
  * Survival (12months, 24 months and at the end of the follow up).
Number of hospitalization during follow up. | 2 years
Evaluation of clotting activator marker with and without Xarelto. | 2 years
Duration of hospitalization during follow up. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Dr Plessier, Principal Investigator — Hôpital Beaujon - APHP
Locations (1):
- Hôpital Beaujon, Clichy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Plessier A, Goria O, Cervoni JP, Ollivier I, Bureau C, Poujol-Robert A, Minello A, Houssel-Debry P, Rautou PE, Payance A, Scoazec G, Bruno O, Corbic M, Durand F, Vilgrain V, Paradis V, Boudaoud L, de Raucourt E, Roy C, Gault N, Valla D. Rivaroxaban Prophylaxis in Noncirrhotic Portal Vein Thrombosis. NEJM Evid. 2022 Dec;1(12):EVIDoa2200104. doi: 10.1056/EVIDoa2200104. Epub 2022 Nov 22. PMID 38319842